CLINICAL TRIAL: NCT00804401
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Two Oral Formulations of Naproxen 500 mg Tablets Administered as 1 x 500 mg Tablet in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study Between Two Oral Formulations of Naproxen 500 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Perrigo Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40061
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Bioequivalency
Keywords: bioequivalency; Naproxen
MeSH Terms: interventions — Naproxen

ARMS (2):
- Test Product (Active Comparator)
  Interventions: Drug: Naproxen Tablets, 500 mg
- Reference Product (Active Comparator)
  Interventions: Drug: Naproxen Tablets, 500 mg

INTERVENTIONS:
Drug: Naproxen Tablets, 500 mg

SUMMARY:
Compare the rate and extent of absorption of two oral formulations of Naproxen Tablets, administered as a 1 x 500 mg tablet under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy men or women, non-smoker, 18 years of age or older
* willing to participate and sign a copy of the informed consent form

Exclusion Criteria:

* clinically significant illnesses or surgery within 4 weeks prior to study dosing
* body mass index greater than or equal to 30.0
* recent history of drug or alcohol addiction or abuse
* pregnant or lactating women
* history of allergic response to naproxen, NSAIDs, or other related drugs, or to heparin
* history of allergic reactions such as asthma, rhinitis, nasal polyps, urticaria, and hypotension associated with the use of aspirin or other NSAIDs
* history or known presence of gastrointestinal ulceration, bleeding and perforation
* use of tobacco products within 6 months prior to study dosing
* evidence of a clinically significant disorder or whose laboratory results were deemed to be clinically significant
* receipt of any drugs as part of a research study within 30 days prior to study dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-06; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence was assessed on the pharmacokinetic variables Cmax, AUC,0-t, and AUC,0-infinity